CLINICAL TRIAL: NCT00684944
Title: An Open Label Continuation Study of the Effects of TRx0014 30 mg TID and 60 mg TID in Patients With Alzheimer's Disease
Brief Title: Open Label Study of TRx0014 in Alzheimer's Disease
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: TauRx Therapeutics Ltd (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: TRx-014-009
Record Dates: First submitted 2008-05-22; First posted 2008-05-28 (Estimated); Last update posted 2018-04-27 (Actual); Status verified 2018-04

CONDITIONS: Alzheimer's Disease
MeSH Terms: conditions — Alzheimer Disease

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- 1 (Active Comparator): 30mg tid TRx0014
  Interventions: Drug: TRx0014
- 2 (Active Comparator): 60mg tid TRx0014
  Interventions: Drug: TRx0014

INTERVENTIONS:
Drug: TRx0014 — Gelatin capsule, tid

SUMMARY:
This is an open label, dose-ranging study of two doses of TRx0014 in patients with mild or moderate Alzheimer's Disease. The trial is made available to any patient ongoing on treatment in the clinical trial designated TRx-014-001 at termination of that study. Treatment for each individual patient will continue for as long as the treating physician feels there is benefit to the patient. This current protocol covers each patient for 12 months in the first instance.

ELIGIBILITY:
Inclusion Criteria:

* The patient may be of either sex and must be supervised by a carer who is competent to ensure compliance with the medication and who is willing to participate in completing the various assessments. The carer must provide written consent to his or her own participation in the study.
* Patients with capacity must give written informed consent to participate in this study. Patients who lack capacity to consent must be in agreement with entering into the study and have a personal legal representative giving written informed consent to their participation.
* The patient must have been ongoing in TRx-014-001 at time of study termination.

Exclusion Criteria:

* There are no exclusion criteria. All patients taking medication at the termination of study TRx-014-001 and who wish to participate are eligible for recruitment.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 111 (Actual)
Dates: Start 2007-09-13 (Actual); Primary Completion 2010-12-02 (Actual); Study Completion 2010-12-02 (Actual)

PRIMARY OUTCOMES:
Cognitive ability measured by the Alzheimer's Disease Assessment Scale - cognitive subscale (ADAS-cog) and by the Mini-Mental State Examination (MMSE). | 0, 26 and 52 weeks

SECONDARY OUTCOMES:
Dementia severity assessed by the Clinical Dementia Rating - sum of the boxes (CDR-sb). | 0, 26 and 52 weeks
Daily living activities assessed by the Alzheimer's Disease functional Assessment and Change Scale (ADFACS) | 0, 26 and 52 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Peter Bentham, MRCPsych, Principal Investigator — Queen Elizabeth Psychiatric Hospital, United Kingdom